CLINICAL TRIAL: NCT05315479
Title: A Phase 4, Multicenter, Open-Label Study to Evaluate the Safety and Pharmacokinetics of N1539 in Children 2 to <17 Years of Age Following Surgery
Brief Title: Safety and Pharmacokinetics of N1539 in Children 2 to <17 Years of Age Following Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Anjeso (N1539) NDA Withdrawn
Sponsor: Baudax Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDX-20-002
Record Dates: First submitted 2022-03-15; First posted 2022-04-07 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Post Operative Pain
Keywords: meloxicam; pediatric
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- N1539 (Experimental): N1539 (Meloxicam IV) 0.6 mg/kg (maximum 30 mg) Q24H
  Interventions: Drug: N1539

INTERVENTIONS:
Drug: N1539 — Once daily
  Other Names: Meloxicam IV

SUMMARY:
This study is an open-label, multicenter evaluation of Safety and Pharmacokinetics of N1539 in postoperative Pediatric subjects aged 2 to <17 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 2 to <17 years of age before dosing on Day 1
* Eligible for elective surgery that will be performed according to standard surgical technique under appropriate anesthesia
* Be premenarche or have confirmed negative urine pregnancy testing before surgery on Day 1, if an adolescent female of childbearing potential
* Willing and able to cooperate with all the requirements of the study; including providing appropriate informed consent/assent

Exclusion Criteria:

* Have a known allergy or hypersensitivity to meloxicam, aspirin, other non-steroidal anti-inflammatory drugs (NSAIDs), or any excipient of N1539
* Have a known bleeding disorder that may be worsened with the administration of an NSAID
* Be undergoing cardiothoracic surgery
* Has used meloxicam within 7 days before the surgical procedure on Day 1
* Has any clinically significant medical history or clinical manifestations of significant disease or any other condition that increases the risk associated with the subject's participation in the study or compromises the scientific objectives of the study.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Center, Sheffield, Alabama
  - Research Center, Bakersfield, California
  - Research Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N1539
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | N1539
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 16 [12 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing an AE
Description: Number of study subjects who experienced an AE
Time Frame: Through study completion, approximately 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | N1539
Number analyzed (Participants) | 19
Participants | 3

ADVERSE EVENTS:
Time Frame: 28 Days following study dosing
Arm/Group | N1539
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 3/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N1539 (N=19)
Tooth infection (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Discussion and/or publication of data generated is not permitted without the prior written consent of the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT05315479/Prot_SAP_002.pdf